CLINICAL TRIAL: NCT06200532
Title: Footwear Self-Assessment Kit for People With Diabetes at Risk of Ulceration - A Feasibility Study
Brief Title: FOOTSAK (Footwear Self-Assessment Kit)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0947
Record Dates: First submitted 2023-12-19; First posted 2024-01-11 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single cohort of people using home footwear self-assessment kit (Experimental): FOOTSAK is a Footwear Self-Assessment Kit intended to empower people with diabetes by providing the necessary tools and instructional materials to enable self-assessment to determine whether footwear has adequate length and width. This feasibility study aims to determine whether people with diabetes and their footwear buddies can use FOOTSAK with sufficient (1) accuracy, (2) reliability and (3) ease of use to identify incorrectly fitting footwear (IFF).
  We will recruit ten people with type 1 or 2 diabetes without any minor or major toe or foot amputation to use the FOOTSAK. Given that foot measurements have to be made whilst standing (to ensure full blood flow to feet during measurements), we will also recruit ten 'Footwear buddies' - people with or without diabetes willing to measure the feet of participating people with diabetes (for example, a spouse, partner, carer, friend, neighbour, or housemate).
  Interventions: Other: FOOTSAK (FOOTwear self-assessment kit)

INTERVENTIONS:
Other: FOOTSAK (FOOTwear self-assessment kit) — FOOTSAK is a Footwear Self-Assessment Kit intended to empower people with diabetes by providing the necessary tools and instructional materials to enable self-assessment to determine whether footwear has adequate length and width. It includes measuring tools (an internal footwear length gauge, scale dividers for measuring internal footwear width, a slide rule for measuring foot length and width, a ruler and magnifying glass for reading off measurements) and instructional materials (booklet instructions and video materials)

SUMMARY:
FOOTSAK is a Footwear Self-Assessment Kit intended to empower people with diabetes by providing the necessary tools and instructional materials to enable self-assessment to determine whether footwear has adequate length and width. This feasibility study aims to determine whether people with diabetes and their footwear buddies can use FOOTSAK with sufficient (1) accuracy, (2) reliability and (3) ease of use to identify incorrectly fitting footwear (IFF).

Ten people with type 1 or 2 diabetes without any minor or major toe or foot amputation will be recruited to use the FOOTSAK. Given that foot measurements have to be made whilst standing (to ensure full blood flow to feet during measurements), ten 'Footwear buddies' - will also be recruited. These are people with or without diabetes willing to measure the feet of participating people with diabetes (for example, a spouse, partner, carer, friend, neighbour, or housemate).

Both participants are asked to watch instructional videos/short demonstrations and read large text instructions. Footwear buddies are asked to repeatedly measure the feet of people with diabetes. People with diabetes are asked to repeatedly measure their footwear then assess whether they are correctly fitting. The feet and footwear of participants with diabetes are then measured by a trained researcher to determine accuracy.

1. Determine whether foot measurements made by footwear buddies are accurate: +/- up to 5mm when compared to a trained researcher.
2. Determine whether repeated footwear and foot measurements made by participants are reliable: Intraclass Correlation Coefficient ≥0.83 for footwear length and ≥0.72 for footwear width (assuming a 15% decrease in reliability when compared to a trained researchers' scores).
3. Determine whether FOOTSAK measuring tools and instructional materials ease of use ≥7.0 /10.0 using Visual Analogue Score with free text comments. Any measuring tool failing to obtain a score of 7.0 or higher will be replaced in consultation with PPI participants and any instructional tool amended through PPI.

ELIGIBILITY:
1. People with type 1 or type 2 diabetes; with or without neuropathy; with or without a history of ulceration who have not had a minor or major amputation;
2. 'Footwear buddies' who consist of people with or without diabetes who are willing to measure the feet of participating people with diabetes - for example, a spouse, partner, carer, friend, neighbour, or housemate.

Inclusion criteria for participant type (1)

1. people who self-report as having type 1 or type 2 diabetes;
2. aged 18 years or over
3. without minor or major amputation
4. Without significant foot deformity
5. Able to read and understand English
6. Willingness and capacity to participate in the study and to sign the informed consent form

Inclusion criteria for participant type (2)

1. Aged 18 or over
2. Willing to act as a 'footwear buddy' for a person with diabetes
3. Able to read and understand English
4. with a willingness and capacity to participate in the study and to sign the informed consent form

Exclusion criteria for participant type (1)

1. Does not self-report as having diabetes (either type 1 or 2)
2. Not aged 18 or over
3. Has minor or major amputation
4. Has significant foot deformity
5. Unable to read and understand English
6. Unwilling or lacking capacity to participate

Exclusion criteria for participant type (2)

1. Not aged 18 or over
2. Unwilling to act as a 'footwear buddy' for a person with diabetes
3. Unable to read and understand English
4. Unwilling or lacking capacity to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Accuracy | Visit 1 on day 1
  Accuracy: average (mean) variation of study participants' foot and footwear measurements from a trained researcher's measurements and standard error of measurements.
Reliability | Visit 1 on day 1
  Intrarater reliability (Intraclass Correlation Coefficient) based on four measurements of the feet and footwear by study participants
Ease of use scores | Visit 1 on day 1
  Mean ease of use visual analogue scores (i) both overall and for each section of instructional material; (ii) for each study video / demonstration and overall; and (iii) both overall and for each measuring tools included within the FOOTSAK

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Research Centre, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Jones PJ, Bullock J, Weaving L, Davies MJ, Razieh C, Ahmad E. Effectiveness of diabetes footwear fit assessment by people with diabetes and their family or partners: A reliability study. Diabet Med. 2025 Aug;42(8):e70065. doi: 10.1111/dme.70065. Epub 2025 Jun 15. PMID 40518605